CLINICAL TRIAL: NCT04758975
Title: Venetoclax and Delayed Rituximab With Ibrutinib Consolidation Aiming at Undetectable Minimal Residual Disease (uMRD) in Treatment-naïve Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Venetoclax, Rituximab and Ibrutinib in TN Patients With CLL Undetectable Minimal Residual Disease (uMRD) in Treatment-naïve Patients With Chronic Lymphocytic Leukemia (CLL)
Acronym: VALUABLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paolo Ghia (Other)
Responsible Party: Sponsor-Investigator, Paolo Ghia, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-CLL-009
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Rituximab +/- Ibrutinib (Experimental): VENETOCLAX: Cycle 1 Day 1-Cycle 1 Day 28 Ramp-up with weekly dose escalation; Cycles 2-12: 400 mg QD RITUXIMAB: Cycle 7 Day 1 375 mg/m2; Cycles 8-12 Day 1 500 mg/m2
  At the end of Cycle 12 the MRD status is checked:
  3 consecutive uMRD in PB + 1 uMRD in BM at last assessment treatment discontinuation and follow-up At least 1 MRD+ sample in the last 3 assessments venetoclax 400 mg QD until uMRD or up to 24 months or unacceptable toxicity (whichever occurs first) in combination with IBRUTINIB 420 mg QD until uMRD or PD or unacceptable toxicity
  Interventions: Drug: Venetoclax; Drug: Rituximab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Venetoclax — VENETOCLAX: Ramp-up than 400 mg QD
Drug: Rituximab — RITUXIMAB: Cycle 7 Day 1 375 mg/m2; Cycles 8-12 Day 1 500 mg/m2
Drug: Ibrutinib — IBRUTINIB 420 mg QD

SUMMARY:
This is a Phase 2, multicenter, open-label uncontrolled interventional study aimed a determining therapeutic benefits of the addition of ibrutinib to 12 months of venetoclax (single-agent for 6 months then combined with rituximab for additional 6 months) in patients with treatment-naïve CLL based on a MRD-guided approach. Study treatment will be administered according to the following scheme:

VENETOCLAX: Cycle 1 Day 1-Cycle 1 Day 28 Ramp-up with weekly dose escalation; Cycles 2-12: 400 mg QD RITUXIMAB: Cycle 7 Day 1 375 mg/m2; Cycles 8-12 Day 1 500 mg/m2

At the end of Cycle 12 the MRD status is checked:

3 consecutive uMRD in PB + 1 uMRD in BM at last assessment treatment discontinuation and follow-up At least 1 MRD+ sample in the last 3 assessments. Venetoclax 400 mg QD until uMRD or up to 24 months or unacceptable toxicity (whichever occurs first) in combination with IBRUTINIB 420 mg QD until uMRD or PD or unacceptable toxicity. Venetoclax will be administered orally once daily (QD) beginning with a dose-titration phase (Ramp-up Period). At Cycle 7 Day 1 rituximab will be added for up to 6 monthly cycles (Cycle 7 Day 1 rituximab 375 mg/m2, Cycles 8-12 Day 1 rituximab 500 mg/m2). At Cycle 12 Day 1, disease status, renal function and risk of bleeding will be assessed. Minimal residual disease (MRD) will be evaluated serially in both PB and, after 3 consecutive uMRD in PB, in BM. All subjects with uMRD (defined as those with MRD level <10-4 in the PB in 3 consecutive assessments and in a BM aspirate) will discontinue venetoclax at the end of Cycle 12 (i.e. Cycle 12 Day 28). All subjects with detectable MRD (defined as those with MRD level in the PB and/or BM >10-4) and patients with stable disease without any contraindications to ibrutinib will start treatment with ibrutinib. Ibrutinib will be administered at the standard dose in CLL (i.e. 420 mg QD). Venetoclax will be administered until confirmed uMRD (3 consecutive uMRD in PB, the last one with concomitant uMRD in BM), unacceptable toxicity or disease progression or for a maximum of 2 years and ibrutinib will be continued until unacceptable toxicity, confirmed uMRD or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years but <65 years
2. Active CLL/SLL requiring treatment per iwCLL 2018 criteria
3. No previous therapy for CLL/SLL
4. Adequate bone marrow function:

   1. ANC ≥1.0 x 109/L;
   2. Plt ≥25 x 109/L;
   3. Hgb ≥8.0 g/dl

Exclusion Criteria:

1. Any prior therapy used for treatment of CLL or SLL
2. History of other malignancies, except in situ carcinoma or malignancy treated with curative intent
3. Known or suspected history of Richter's transformation
4. Known hypersensitivity to one or more study drugs
5. Inadequate renal function: CrCl <30 mL/min
6. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
7. Requires the use of warfarin or derivatives
8. Treatment with any of the following within 7 days prior to the first dose of study drug:

   1. Steroid therapy for anti-neoplastic intent
   2. Moderate or strong cytochrome P450 3A (CYP3A) inhibitors (see Appendix G for examples)
   3. Moderate or strong CYP3A inducers (see Appendix G for examples)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
uMRD (<10-4) by 6-color flow cytometry in the bone marrow | 27 months
  uMRD (<10-4) by 6-color flow cytometry in the bone marrow as best response at any time during treatment for up to 3 months after completion of combined therapy (VR or VR followed by VI)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No